CLINICAL TRIAL: NCT02052973
Title: Efficacy of Brazilian Green Propolis Varnish Against Streptococcus Mutans in Saliva: a Phase II Study.
Brief Title: Efficacy of Propolis Varnish Against Oral Biofilm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Mariana Passos De Luca, DDS, MSc, PhD student, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10726612.8.0000.5149
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Streptococcal Infections; Saliva Altered
Keywords: Streptococcus mutans; Natural products
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propolis varnish (Experimental): Saliva and oral biofilm will be collected before and in regular times after the application of the propolis varnish. This data will be compared in order to evaluate the probable reduction of Streptococcus mutans in saliva and oral biofilm.
  Interventions: Other: Propolis varnish

INTERVENTIONS:
Other: Propolis varnish — Saliva and oral biofilm will be collected before and in regular times after the application of the propolis varnish. This data will be compared in order to evaluate the probable reduction of Streptococcus mutans in saliva and oral biofilm.

SUMMARY:
This study aims to evaluate the effectiveness of a varnish containing 15% of green propolis on Streptococcus mutans in saliva and biofilm. Will be invited to join the study: children 8-10 years old, free of caries, without orthodontic appliances and without having undergone antibiotic therapy until three weeks before the start of the study. Saliva will be collected before, immediately after, 24 hours and 30 days after application of the varnish. The collection of biofilm will be performed before, after, 24 hours and 30 days after application of the varnish. Data will be collected and compared between periods.

DETAILED DESCRIPTION:
Antimicrobials are substances used in dentistry as an efficient way of caries prevention. Substances such as chlorhexidine are the most known and most applied for this purpose and, as a varnish, increased its anticariogenic potential. The antimicrobial effects of natural substances are being studied for exhibiting antimicrobial properties similar to those of chlorhexidine, but less toxic in some cases. Several studies with propolis has proven its efficacy against several microorganisms of the oral cavity, specially Streptococcus mutans. A pharmaceutical formulation containing brazilian green propolis was developed based on the chitosan polymer that is biocompatible and biodegradable. In a previous study, we observed in vitro antimicrobial properties of the varnish against Streptococcus mutans. This work aims to study the preliminary evidence of the efficacy of the propolis dental varnish in reducing Streptococcus mutans in saliva and in the biofilm control through a phase II study involving patients with 8-10 years. After 30 days, the results will be compared and statistically analyzed at a level of significance of 5 % .

ELIGIBILITY:
Inclusion Criteria:

* children 8-10 years old
* good general health condition
* not making use of mouthwashes or medications (especially antibiotics), until three weeks prior to the beginning of the experiment.

Exclusion Criteria:

* Patients in medical treatment or who used drugs (especially antibiotics), in the three previous weeks and patients with active caries lesions.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Streptococcus mutans in saliva and in tooth biofilm | 30 days

SECONDARY OUTCOMES:
Caries incidence reduction | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariana P De Luca, DDs MSc, Principal Investigator — UFMG